CLINICAL TRIAL: NCT01320618
Title: Prospective Cohort Study of Robotic Assisted Laparoscopic Sacrocolpopexy Using MPATHY Restorelle Mesh
Acronym: MPATHY
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, Principal Investigator, Atlantic Health System
Other Study IDs: R09-06-003
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Organ Prolapse; Urinary Incontinence; Mesh Erosion
Keywords: uterine prolapse; vaginal prolapse; mesh erosion; urinary incontinence; bowel symptoms
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence; Uterine Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Robotic approach to sacral colpopexy is a relatively new procedure. The literature is scarce in regard to long term outcome. This advanced procedure is offered at Morristown Memorial. This protocol will review the one year outcome of patients who underwent this procedure using a polypropylene mesh. These outcomes will include anatomical and quality of life measures.

ELIGIBILITY:
Inclusion Criteria:

* Any patient receiving Robotic assisted laparoscopic sacral colpopexy with polypropylene mesh

Exclusion Criteria:

* Other graft material than polypropylene mesh
* Enrollment in another study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study population will be woman who underwent Robotic assisted laparoscopic sacral colpopexy at the Morristown Memorial Hospital for correction of pelvic organ prolapseusing synthetic polypropelene mesh.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)